CLINICAL TRIAL: NCT07041359
Title: Pre-trial of Clinical Trial of Traditional Chinese Medicine Treatment for Elderly Patients With Coronary Heart Disease Who Are Still Symptomatic After Optimal Medical Treatment
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-ZX080
Record Dates: First submitted 2025-06-06; First posted 2025-06-27 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-02

CONDITIONS: Coronary Arterial Disease (CAD)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Qi stagnation and blood stasis type control group (Placebo Comparator): Intervention with placebo on the Basis of optimal medical treatment
  Interventions: Drug: Placebo
- Qi stagnation and blood stasis type experimental group (Experimental): Intervention with Compound Danshen Dripping Pills on the Basis of optimal medical treatment
  Interventions: Drug: Compound Danshen Dripping Pills
- Qi deficiency and blood stasis type control group (Placebo Comparator): Intervention with placebo on the Basis of optimal medical treatment
  Interventions: Drug: Placebo
- Qi deficiency and blood stasis type experimental group (Experimental): Intervention with Qishen Yiqi Dropping Pills on the basis of conventional western medicine treatment
  Interventions: Drug: Qishen Yiqi Drop Pills

INTERVENTIONS:
Drug: Compound Danshen Dripping Pills — The experimental group used compound Danshen dripping pills as an intervention on the basis of conventional western medicine treatment.
  Arms: Qi stagnation and blood stasis type experimental group
Drug: Qishen Yiqi Drop Pills — The experimental group used Qishen Yiqi dripping pills as an intervention on the basis of conventional western medicine treatment.
  Arms: Qi deficiency and blood stasis type experimental group
Drug: Placebo — Intervention with placebo on the Basis of optimal medical treatment
  Arms: Qi deficiency and blood stasis type control group; Qi stagnation and blood stasis type control group

SUMMARY:
To explore the effectiveness of compound Danshen Dripping Pill and Qishen Yiqi Dripping Pill in the elderly population with coronary heart disease and the safety of multiple medications

DETAILED DESCRIPTION:
This study is a prospective, double-blind, randomized controlled clinical trial, which aims to explore the effectiveness and safety of polypharmacy in the elderly population of stable angina patients, and make up for the limitations of clinical treatment. As commonly used traditional Chinese medicine preparations, the efficacy and safety of compound Danshen Dripping Pill and Qishen Yiqi Dripping Pill have been supported by previous studies, providing a solid theoretical basis. The study design adopts scientific and reliable clinical trial methods, and the treatment plan combines Western medicine treatment and traditional Chinese medicine intervention, which has high clinical application value. In the actual clinical treatment, due to the complex medical history of elderly patients, they often have multi-vessel coronary artery lesions, and the treatment tolerance is worse than that of young people, so although they are accompanied by angina pectoris, the treatment methods are relatively limited. This study provides evidence of the efficacy and safety of drugs for the treatment of elderly patients with angina pectoris through the combination of Chinese and Western treatments, which can help make up for the dilemma of limited clinical treatment methods.

ELIGIBILITY:
Inclusion Criteria:

1. 75 years old ≤ age < 90 years old, regardless of gender;
2. Patients who meet the diagnostic criteria for angina pectoris, including patients with typical or atypical angina pectoris: discomfort in the anterior region is triggered by physical activity or emotional excitement and can be relieved by rest or taking nitroglycerin.Those who meet two or more of the above characteristics. After receiving conventional Western medicine treatment, the symptoms did not improve significantly or the treatment effect is poor.
3. Meet the diagnostic criteria for multiple coronary artery disease with the number of coronary artery disease being greater than or equal to two (defined as angiographically the right coronary artery, left circumflex artery or left anterior descending artery stenosis rate was greater than 50%), and the patient refused or could not tolerate coronary artery revascularization or one or more coronary arteries still have a stenosis rate of ≥50% after partial revascularization;
4. The patient is in line with the qi stagnation and blood stasis type or qi deficiency and blood stasis type in the TCM syndrome classification. If the results of the two syndrome differentiation are inconsistent, the TCM experts will review the syndrome differentiation, and the syndrome differentiation classification of the TCM experts shall prevail.
5. The patient has good communication skills, can understand and provide relevant information required for the study, and is aware of the research purpose, content, possible risks and expected benefits can be fully provided with relevant information required for this research. Patients and their families voluntarily participated and agreed to sign the informed consent.

Exclusion Criteria:

1. Those who have had acute coronary syndrome within the past month
2. Acute myocardial infarction, acute myocarditis, severe arrhythmia, aortic dissecction, pericarditis, heart failure (NYHA heart function class Ⅲ or IV, EF ≤ 30%), cardiogenic shock in past 3 months or patients with chest tightness and chest pain caused by other diseases such as severe valvular disease, etc.
3. Combined with acute pulmonary embolism, acute cerebral hemorrhage, polyarteritis, severe hematologic diseases, severe infectious diseases, severe immune dysfunction, malignant tumors, other organ failure or expected life expectancy less than 1 year
4. Severe primary disease or severe dysfunction of the liver or kidneys（ALT levels exceeding 3.0 times the upper limit of normal or eGFR ≤30 mL/min/1.73 m²）
5. Patients with severe mental disorder
6. Those who are allergic to the test drug
7. Patients who have participated in other clinical trials in the past month
8. Patients who have taken anticoagulants such as warfarin, new oral anticoagulants (NOAC) or traditional Chinese medicine preparations for promoting blood circulation and removing blood stasis in the past month
9. Refusal to sign informed consent

Ages: 75 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Seattle angina questionnaire | 8 weeks. If the change is not significant, it can be extended to 12 weeks.
  The Seattle Angina Questionnaire (SAQ) consists of five distinct dimensions: physical limitation, angina stability, angina frequency, treatment satisfaction, and disease perception. Each dimension is scored independently, with a possible range of 0 to 100 points. A higher score on any SAQ dimension indicates a better patient condition or experience.
The Canadian Cardiovascular Society grading of angina pectoris | 8 weeks. If the change is not significant, it can be extended to 12 weeks.
  The Canadian Cardiovascular Society grades angina pectoris ranges from grade 1 to grade 4. Higher grade indicates worse patients' condition.
Minnesota Living with Heart Failure Questionnaire | 8 weeks. If the change is not significant, it can be extended to 12 weeks.
  The Minnesota Living with Heart Failure Questionnaire's score ranges from 0 to 105. Higher score indicates worse patients' condition.
Kansas City Cardiomyopathy Questionnaire | 8 weeks. If the change is not significant, it can be extended to 12 weeks.
  The Kansas City Cardiomyopathy Questionnaire's score ranges from 0 to 100. Higher score indicates better patients' condition.

SECONDARY OUTCOMES:
Traditional Chinese Medicine Syndrome Score | 8 weeks. If the change is not significant, it can be extended to 12 weeks.
  The Traditional Chinese Medicine Syndrome Score ranges from 0 to 30. Higher score indicates worse patients' condition.
Number of angina attacks | 8 weeks. If the change is not significant, it can be extended to 12 weeks.
  The average number of angina attacks per week
Nitroglycerin dosage | 8 weeks. If the change is not significant, it can be extended to 12 weeks.
  Patient's weekly dose of nitroglycerin, measured in mg

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai hospital, CAMS&PUMC, Beijing, Beijing Municipality, China